CLINICAL TRIAL: NCT07360366
Title: Interprofessional Collaboration in the Cardiac Intensive Care Unit (CICU): An Action-Research Training Project
Acronym: COLLUTIC_25
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Santina Gavagni, Nurse, Azienda Ospedaliero-Universitaria di Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 502/2025/OSS /AOUPR
Record Dates: First submitted 2025-12-31; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Interprofessional Relations; Interprofessional Education; Attitude of Health Personnel; Intensive Care Units; Critical Care
Keywords: Interprofessional Relations; Interdisciplinary Communication; Health Personnel Attitudes; Nurse-Physician Relations; Intensive Care Units; Coronary Care Units; Critical Care; Patient Care Team; Education, Interprofessional; Clinical Decision-Making
MeSH Terms: interventions — Physicians; Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental): The training phase of the project consists of an interactive course aimed at healthcare professionals (physicians, nurses and OSS) to improve their ability to recognise and enact effective collaborative practices. Learning is based on the use of branching scenarios, created with the H5P software. This approach enables learners to distinguish correct practices and refine their teamwork skills. The course also provides access to additional content on techniques and procedures specific to the UTIC context, curated by expert professionals.
  Interventions: Other: The training phase of the project consists of an interactive course aimed at healthcare professionals (physicians, nurses and OSS) to improve their ability to recognise and enact effective collaborati

INTERVENTIONS:
Other: The training phase of the project consists of an interactive course aimed at healthcare professionals (physicians, nurses and OSS) to improve their ability to recognise and enact effective collaborati — The branching scenarios replicate complex and common clinical situations that require effective interprofessional collaboration. Each scenario is carefully designed with detailed clinical and organisational elements, including the simulated patient's medical history and care pathway in the cath-lab and electrophysiology unit prior to a TAVI procedure, vital signs, diagnostic tests, available resources, clinical objectives, and potential critical issues. Scenarios are structured around a defined storyline and professional roles, and are divided into key phases with information, possible actions, and related consequences. Interactive elements allow learners to make decisions and engage with characters or objects, while meaningful feedback supports learning. Multiple pathways ensure a dynamic experience, supported by assessment criteria.

SUMMARY:
This study evaluates the impact of a structured interprofessional training program on daily collaboration within the Cardiac Intensive Care Unit (CICU/UTIC) at the University Hospital of Parma. In high-intensity clinical settings, rapid and accurate coordination between physicians, nurses, and healthcare assistants is vital. Ineffective teamwork often leads to communication breakdowns, potentially compromising patient safety and care quality. This project investigates whether an interactive, scenario-based educational program can strengthen role clarity, communication, and shared decision-making.

The study seeks to determine if an active-learning program using interactive branching scenarios improves interprofessional collaboration more effectively than traditional methods. The researchers hypothesize that this simulation-based approach will significantly enhance professional outcomes, including self-efficacy, shared decision-making, and commitment to both the team and the profession.

The study utilizes a convenience sample (approx. 5 physicians, 30 nurses, 8 healthcare assistants, and 10 students). Eligible participants include staff and students currently or recently active in the Parma CICU who provide informed consent.

The intervention is delivered via a Moodle-based platform featuring case-based simulations. These scenarios replicate complex clinical pathways, such as:

Cath-lab and Electrophysiology procedures.

Heart failure management.

TAVI (Transcatheter Aortic Valve Implantation) preparation.

As participants navigate these scenarios, they must make critical decisions and receive immediate feedback designed to reinforce collaborative best practices.

Data Collection and Timeline

Data is gathered at three intervals: T0 (Baseline), T1 (Post-training), and T2 (6-month follow-up). Validated questionnaires measure:

Attitudes toward physician-nurse collaboration.

Perceived daily collaboration and decision-making satisfaction.

Professional commitment and work-related self-efficacy.

The training phase spans six months, with a subsequent six-month follow-up, totaling a 24-month project duration.

Ethics and Privacy Risks are minimal, primarily involving the time required for participation. The primary benefit is the development of skills that foster safer, more coordinated patient care. Privacy is strictly maintained through pseudo-anonymization, with data access restricted to the research team.

DETAILED DESCRIPTION:
Background and Rationale Interprofessional collaboration is critical for patient safety and organizational efficiency in high-complexity environments like the Cardiac Intensive Care Unit (CICU). Despite its importance, there is a lack of structured, transferable training models for daily clinical practice. Poor cooperation is linked to preventable adverse events and caregiver burnout. This study, promoted by the Azienda Ospedaliero-Universitaria di Parma, addresses this gap using an "action-research" approach integrated with digital tools for situated learning.

Study Design and Intervention This is a longitudinal, prospective study. The intervention consists of a specialized training program using interactive branching scenarios created with H5P software and hosted on a Moodle-based platform. These simulations replicate complex clinical situations across four key CICU pathways:

Hemodynamics. Electrophysiology. Heart Failure. TAVI (Transcatheter Aortic Valve Implantation) preparation. The program requires learners to make clinical and collaborative decisions, receiving immediate feedback to improve teamwork, role clarity, and communication.

Data Collection and Analysis The study evaluates outcomes at three specific intervals:

T0: Baseline (pre-intervention). T1: Post-intervention (immediately following training). T2: Follow-up at six months to evaluate sustainability Assessment tools include the Jefferson Scale of Attitudes Toward Physician-Nurse Collaborative Relationship (JSAPNC) , the Nurse-Physician Collaboration Scale (NPCS) , and the Maslach Burnout Inventory (MBI) for self-efficacy. Statistical evaluation will utilize Linear Mixed Models (LMM) to analyze longitudinal changes and individual trajectories.Ethics and Data Management The study follows a pseudo-anonymized data protocol, with access restricted to the research team. Participants provide written informed consent prior to enrollment. The project duration is estimated at 24 months.

The study is projected to commence on February 15, 2026.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals (physicians, nurses and healthcare assistants/OSS) employed in the Cardiac Intensive Care Unit (UTIC) of the University Hospital of Parma.
* Healthcare professionals who have completed the training pathway and are still working in the unit at the time of the six-month follow-up.
* Medical and nursing students who have carried out or are carrying out a clinical placement within the UTIC.
* Ability to use a computer or mobile device, essential for participating in the online training activities (e.g. Moodle, H5P).
* Provision of written informed consent before initiation of any study procedure.

Exclusion Criteria:

* Healthcare professionals who do not work in the cardiology setting or who are not employed in the UTIC of the AOU Parma.
* Inability to participate in the training activities or assessment sessions for logistical, organisational or clinical reasons (e.g. planned prolonged absences during the study period).
* Refusal or inability to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Name of the measurement: Change from Baseline in Mean Attitudes Toward Physician-Nurse Interprofessional Collaboration Score at 6 Months | Baseline (T0), immediately post-training (T1: approximately 1 month after baseline), and at 6-month follow-up (T2: 6 months after the intervention).
  Measurement tool: Jefferson Scale of Attitudes Toward Physician-Nurse Collaborative Relationship (JSAPNC); Unit of measure: Mean total score on the Jefferson Scale of Attitudes toward Physician-Nurse Collaboration;Attitudes toward physician-nurse interprofessional collaboration will be assessed using JSAPNC, a structured, self-administered questionnaire designed to evaluate attitudes toward collaborative relationships between physicians and nurses. JSAPNC assesses key aspects of physician-nurse collaboration, including mutual respect, shared responsibility, teamwork, and professional roles. Participants respond to a series of items using a standardized response scale, and item responses are combined to generate a total score representing overall attitudes toward physician-nurse interprofessional collaboration. Higher total scores indicate more positive attitudes toward collaboration. The outcome measure is defined as the change in mean JSAPNC total score from baseline to 6 months.
Name of the measurement: Change from Baseline in Mean Perceived Interprofessional Collaboration Score at 6 Months as Assessed by the Nurse-Physician Collaboration Scale (NPCS) | T0 (Baseline): Before the start of the training intervention. T1 (Post-intervention): Immediately following the completion of the 6-month training program. T2 (Follow-up): Six months after the conclusion of the training to evaluate the sustainability
  Measurement tool: Nurse-Physician Collaboration Scale (NPCS).Unit of measure: Mean total score on the Nurse-Physician Collaboration Scale (NPCS). Perceived interprofessional collaboration will be assessed using the Nurse-Physician Collaboration Scale (NPCS), a structured, self-administered questionnaire designed to evaluate nurses' and physicians' perceptions of interprofessional collaboration. The NPCS assesses key dimensions of nurse-physician collaboration, including communication, shared decision-making, coordination of care, and professional relationships. Participants respond to a series of items using a standardized response scale, and item responses are combined to generate a total score representing the overall level of perceived interprofessional collaboration. Higher total scores indicate greater perceived collaboration. The outcome measure is defined as the change in mean NPCS total score from baseline to 6 months.
Name of the measurement:Change from Baseline in Mean Collaboration and Satisfaction with Care Decisions (CSACD) Score at 6 Months. Measurement tool: Collaboration and Satisfaction with Care Decisions (CSACD) Scale | T0: Baseline (before the training intervention). T1: Post-intervention (immediately following the 6-month training period). T2: Long-term follow-up (6 months after completing the training).
  Unit of measure: Mean total score on the Collaboration and Satisfaction with Care Decisions (CSACD) scale.
  Perceived collaboration and satisfaction with care decisions will be assessed using the Collaboration and Satisfaction with Care Decisions (CSACD) Scale, a validated, structured, self-administered questionnaire. The CSACD includes 9 items, with a Collaboration subscale (7 items) and a Satisfaction subscale (2 items), rated on a 7-point Likert scale. Item responses are combined to generate a total score representing overall perceived collaboration and satisfaction with care decisions. The outcome measure is defined as the change in mean CSACD total score from baseline to 6 months.
Name of the measurement: Change from Baseline in Mean Professional and Team Commitment Scores at 6 Months as Assessed by the Professional and Team Commitment Questionnaire. Tool measurement: Professional and Team Commitment Questionnaire | T0: Baseline (prior to the training intervention). T1: Post-intervention (immediately following the 6-month training period). T2: Follow-up (6 months after the completion of the training).
  Unit of measure: Mean subscale scores on the Professional Commitment scale (12 items; range 12-60) and the Team Commitment scale (5 items; range 5-25). Professional and team commitment will be assessed using the Professional and Team Commitment Questionnaire, a structured, self-administered questionnaire designed to evaluate levels of commitment to one's profession and to the interprofessional team. The questionnaire assesses key dimensions of professional and team commitment, including identification with professional roles, engagement in team activities, and commitment to collaborative work. Participants respond to a series of items using a standardized response scale, and item responses are combined to generate a total score representing overall professional and team commitment. Higher total scores indicate greater levels of professional and team commitment. The outcome measure is defined as the change in mean Professional and Team Commitment total score from baseline to 6 months.
Name of the measurement: Change from Baseline in Mean Work-related Self-Efficacy Score at 6 Months as Assessed by the Personal Accomplishment Subscale of the MBI Measurement tool: Maslach Burnout Inventory (MBI) - Personal Accomplishment Subscale | Baseline (T0), immediately post-training (T1: ~1 month), and 6-month follow-up (T2).
  Unit of measure: Mean score on the Personal Accomplishment subscale of the Maslach Burnout Inventory (MBI).
  Work-related self-efficacy will be assessed using the Personal Accomplishment Subscale of the Maslach Burnout Inventory (MBI), a structured, self-administered questionnaire designed to evaluate individuals' feelings of competence and achievement in their professional work. The Personal Accomplishment Subscale measures key aspects of work-related self-efficacy, including perceived effectiveness, accomplishment, and competence in performing job-related tasks. Participants respond to a series of items using a standardized response scale, and item responses are combined to generate a total subscale score representing overall work-related self-efficacy. Higher scores indicate greater work-related self-efficacy. The outcome measure is defined as the change in mean Personal Accomplishment subscale score from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Santina Gavagni Principal Investigator, Principal Investigator — Parma University Hospital
Locations (1):
- Parma University Hospital, Parma, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-09-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT07360366/Prot_000.pdf